CLINICAL TRIAL: NCT07264673
Title: A Randomized Phase II Trial of Cemiplimab Plus OSE2101 ( TEDOPI®) as Maintenance Therapy in ctDNA Positive NSCL. The Cemited Study.
Acronym: Cemited
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEMITED
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: NSCLC
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: phase II randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Cemiplimab 350 mg iv q21 single agent (squamous histology) or Cemiplimab 350 mg iv q21 plus pemetrexed 500mg/m2 q21 (non- squamous histology).
  Interventions: Drug: Cemiplimab
- B (Experimental): Cemiplimab 350 mg iv q 21 plus OSE2101 (TEDOPI®). The OSE2101 (TEDOPI®) dose to be injected is of 1 mL (5 mg of drug product) by subcutaneousubcutaneous administration
  Interventions: Drug: Tedopi

INTERVENTIONS:
Drug: Tedopi — Cemiplimab + OSE2101 (TEDOPI®) (ARM B: experimental arm)
  Other Names: Cemiplimab
  Arms: B
Drug: Cemiplimab — Cemiplimab +/-Pemetrexed (ARM A: standard arm)
  Arms: A

SUMMARY:
This is a phase II randomized study investigating whether a combination maintenance with Cemiplimab and OSE2101 (TEDOPI®) could increase ctDNA clearance rate versus standard maintenance therapy in HLA-A2 positive NSCLC patients not progressing after 4 cycles of chemo-immunotherapy.

DETAILED DESCRIPTION:
This is a phase II randomized study investigating whether a combination maintenance with Cemiplimab and OSE2101 (TEDOPI®) could increase ctDNA clearance rate versus standard maintenance therapy in HLA-A2 positive NSCLC patients not progressing after 4 cycles of chemo-immunotherapy.

NSCLC patients with any histology, irrespective of PD-L1 expression levels and candidates for first line metastatic therapy will be screened for HLA-A2 status.

After evaluation of all inclusion and exclusion criteria and after informed consent signature, all eligible patients will receive up to four cycles of chemotherapy and Cemiplimab. The chemotherapy regimen will be selected by the investigator, in accordance with current clinical practice, favoring the use of platinum-based chemotherapy agents.

Patients not progressing after 4 cycles of chemo-immunotherapy will be evaluated for the cTDNA presence (baseline).

If they are positive for ctDNA will be further randomized to standard maintenance therapy or to the combination maintenance of Cemiplimab and OSE2101 (TEDOPI®). In case of ctDNA negative test will be treated with Cemiplimab according to clinical practice.

ctDNA will be further evaluated before cycle 3, and at the time of disease progression or at the end of maintenance therapy.

To summarize ctDNA will be analyzed in patients not progressing after 4 cycles of chemo-immunotherapy (before randomization), during the maintenance therapy and at the time of progression.

An additional blood sample will be collected in all patients at the time of starting first-line chemo-immunotherapy (pre-baseline).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of non- oncogene addicted advanced, locally advanced (not suitable for definitive chemoradiation therapy) or metastatic non-small-cell lung cancer (NSCLC)
* Any patient candidate for first line chemo-immunotherapy irrespective of PD-L1 levels
* HLA-A2 positive
* ECOG PS 0-1
* Signed informed consent (IC) prior to any trial-specific procedures

Exclusion Criteria:

* Patients not candidate for chemo-immunotherapy
* HLA-A2 negative
* Symptomatic or not previously treated and not stable brain metastases. Brain metastases are allowed if asymptomatic or pretreated
* Tumor tissue not available (archive or collected before trial inclusion)
* Evidence of EGFR mutations or ALK or ROS1 rearrangements
* Performance status >1 (ECOG)
* Diagnosis of another cancer in the last 3 years, except for in situ carcinoma of cervix, breast and bladder or skin carcinoma(squamous or basaloid)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance rate | 48 months
  Differences in ctDNA clearance rate in the two arms of treatment
  Differences in ctDNA clearance rate in the two arms of treatment
  Differences in ctDNA clearance rate in the two arms of treatment
  Differences in ctDNA clearance rate in the two arms of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Fisioterapici Ospitalieri- Ifo - Istituto Regina Elena, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided